CLINICAL TRIAL: NCT00135980
Title: Integrated Care for Cancer Patients
Brief Title: Integrated Care for Cancer Patients; Developing, Implementing and Testing a Programme to Improve Integrated Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: PACT-study M2100; M2100
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Behavioral: professional audit and feedback
Behavioral: integrated care programmes

SUMMARY:
The purpose of this study is to compose, implement and evaluate a programme to improve the quality of integrated care for patients with cancer.

Literature will be searched for components of integrated care programmes. On the basis of evidence based multi-disciplinary guidelines and literature on integrated care programmes, a set of indicators will be composed. This set will be measured in 6 hospitals on patients with non-small-cell-lung cancer. In two hospitals, an integrated care programme will be implemented and effects on processes and outcomes of care will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Each new patient that visits the lung specialist in 6 hospitals in the east part of Holland, in the period from September 2004 till March 2005

Exclusion Criteria:

* Mortality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-08; Study Completion 2007-07

PRIMARY OUTCOMES:
guideline adherence

SECONDARY OUTCOMES:
hospitalization
satisfaction
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Rosella Hermens, MSc,PhD, Principal Investigator — Centre for Quality of Care Research, Radboud University Nijmegen Medical Centre; Hub Wollersheim, MD,PhD, Study Director — Centre for Quality of Care Research, Radboud University Medical Centre
Locations (6):
- Netherlands (6):
  - Rijnstate Hospital, Arnhem
  - MaasHospital Pantein, Boxmeer
  - Slingeland Hosptital, Doetinchem
  - Gelderse Vallei Hospital, Ede
  - CWZ Hospital, Nijmegen
  - Radboud University Medical Centre, Nijmegen

REFERENCES:
- [Background] Ouwens M, Wollersheim H, Hermens R, Hulscher M, Grol R. Integrated care programmes for chronically ill patients: a review of systematic reviews. Int J Qual Health Care. 2005 Apr;17(2):141-6. doi: 10.1093/intqhc/mzi016. Epub 2005 Jan 21. PMID 15665066
- See also: Site of the Centre for Quality of Care Research — http://www.wokresearch.nl